CLINICAL TRIAL: NCT04094246
Title: The Effect of Battlefield Acupuncture and Physical Therapy Versus Physical Therapy Alone Following Shoulder Surgery: A Randomized Clinical Trial
Brief Title: Battlefield Acupuncture Following Shoulder Surgery
Acronym: BFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Crowell, Director & Associate Professor, Keller Army Community Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19KACH003
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Shoulder Injuries; Pain, Postoperative; Acupuncture, Ear; Pain Management
MeSH Terms: conditions — Shoulder Injuries; Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in the experimental group will receive standard post-surgical rehabilitation protocol per their surgery in addition to Battlefield Acupuncture.
  Interventions: Procedure: Battlefield Acupuncture
- Control Group (Active Comparator): Participants in the control group will receive standard post-surgical rehabilitation protocol per their surgery.
  Interventions: Procedure: Standard post-surgical rehabilitation

INTERVENTIONS:
Procedure: Battlefield Acupuncture — Battlefield Acupuncture (BFA), an auricular acupuncture protocol developed in 2001 by Dr. Niemtzow (Ret. Colonel, USAF), is widely used among civilian and military medical providers to treat pain. Participants in the Experimental Group will receive BFA in addition to standard post-surgical rehabilitation up to four times following their shoulder surgery: 24-hours, 48-hours, 72-hours, and 1-week post-surgery.
  Arms: Experimental Group
Procedure: Standard post-surgical rehabilitation — Participants will receive rehabilitation and will perform a home exercise program in accordance with the standard post-operative shoulder protocol. Participants will be asked to record compliance on an exercise log.
  Arms: Control Group

SUMMARY:
The purpose of this randomized clinical trial is to determine the effectiveness of Battlefield Acupuncture (BFA) in addition to standard post-surgical shoulder physical therapy compared to a standard shoulder rehabilitation program in reducing medication use and pain in patients who have undergone shoulder surgery. Measurements of medication (opioid, NSAID, acetaminophen, etc.) use (daily number of pills consumed), pain rating, patient specific functional scale and global rating of change will be taken at 48-hours (baseline), 72-hours, 1-week, and 4-weeks post-surgery. It is hypothesized that the inclusion of Battlefield Acupuncture will result in a decrease in post-surgical pain levels, reduced opioid medication use, and improved patient mood when compared to rehabilitation alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 17-55 Department of Defense beneficiaries (17 only if an emancipated cadet at the U.S. Military Academy)
* Prior to or within 48 hours post shoulder stabilization surgery
* Prior to or within 48 hours post rotator cuff repair surgery

Exclusion Criteria:

* Self-reported pregnancy
* History of blood borne pathogens, infectious disease, or active infection
* History of metal allergy
* History of bleeding disorders or currently taking anti-coagulant medications
* Participants who are not fluent in English

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Worst overall pain assessed by Visual Analogue Scale (VAS) | 72 hours, 1 week
  Worst pain intensity in the past 24 hours recorded using a 0-10 cm visual analog scale where 0 equals no pain and 10 indicates the most severe pain the patient could imagine. Higher numbers equal greater levels of reported pain.
Average 24-hour pain assessed by Visual Analogue Scale (VAS) | 72 hours, 1 week
  Average pain intensity in the past 24 hours recorded using a 0-10 cm visual analog scale where 0 equals no pain and 10 indicates the most severe pain the patient could imagine. Higher numbers equal greater levels of reported pain.

SECONDARY OUTCOMES:
Patient self-reported mood assessed by the Profile of Mood States (POMS) Questionnaire | 72 hours, 1 week, 4 weeks
  The POMS consists of 65 measures of mood organized into 6 mood scales: tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue-inertia, and confusion-bewilderment. Individual scales are combined to achieve the mood disturbance score (MDS), an aggregate indicator of overall mood. A greater MDS value indicates greater mood disturbance.
Medication Use | 1 week, 4 weeks
  Daily opioid, NSAID, and Acetaminophen use
Worst overall pain and average pain in the past 24 hours assessed by Visual Analogue Scale (VAS) | 4 weeks
  Worst pain intensity and average pain intensity in the past 24 hours recorded using a 0-10 cm visual analog scale where 0 equals no pain and 10 indicates the most severe pain the patient could imagine. Higher numbers equal greater levels of reported pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Keller Army Community Hospital - Arvin Physical Therapy, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crowell MS, Florkiewicz EM, Morris JB, Mason JS, Pitt W, Benedict T, Cameron KL, Goss DL. Battlefield Acupuncture Does Not Provide Additional Improvement in Pain When Combined With Standard Physical Therapy After Shoulder Surgery: A Randomized Clinical Trial. Mil Med. 2025 Jun 30;190(7-8):e1509-e1517. doi: 10.1093/milmed/usae577. PMID 39797512
- [Derived] Crowell MS, Brindle RA, Mason JS, Pitt W, Miller EM, Posner MA, Cameron KL, Goss DL. The effectiveness of battlefield acupuncture in addition to standard physical therapy treatment after shoulder surgery: a protocol for a randomized clinical trial. Trials. 2020 Dec 3;21(1):995. doi: 10.1186/s13063-020-04909-8. PMID 33272311

DOCUMENTS (1):
  • Informed Consent Form (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT04094246/ICF_000.pdf